CLINICAL TRIAL: NCT02965833
Title: Clinical Study of CLEAR CARE® PLUS for Presbyopic Contact Lens Wearers
Brief Title: CLEAR CARE® PLUS for Presbyopic Contact Lens Wearers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alcon, a Novartis Company (Industry)
Responsible Party: Sponsor
Organization: Alcon Research (Industry)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Supportive Care
Other Study IDs: LCS739-P001
Record Dates: First submitted 2016-11-15; First posted 2016-11-17 (Estimated); Results first posted 2018-04-26 (Actual); Last update posted 2018-07-11 (Actual); Status verified 2018-06

CONDITIONS: Presbyopia
Keywords: Contact lens induced dryness
MeSH Terms: conditions — Presbyopia

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- CCP, then HMPS (Other): 3% hydrogen peroxide solution with HydraGlyde® Moisture Matrix contact lens solution in Period 1, followed by subject's habitual multi-purpose contact lens solution (HMPS) in Period 2. Each product used daily per packaging instructions with subject's habitual contact lenses for approximately 30 cleaning and disinfection cycles.
  Interventions: Device: 3% hydrogen peroxide solution with HydraGlyde® Moisture Matrix; Device: Habitual Multi-Purpose Contact Lens Solution; Device: Habitual Contact Lenses
- HMPS, then CCP (Other): Subject's habitual multi-purpose contact lens solution in Period 1, followed by 3% hydrogen peroxide solution with HydraGlyde® Moisture Matrix contact lens solution in Period 2. Each product used daily per packaging instructions with subject's habitual contact lenses for approximately 30 cleaning and disinfection cycles.
  Interventions: Device: 3% hydrogen peroxide solution with HydraGlyde® Moisture Matrix; Device: Habitual Multi-Purpose Contact Lens Solution; Device: Habitual Contact Lenses

INTERVENTIONS:
Device: 3% hydrogen peroxide solution with HydraGlyde® Moisture Matrix — For cleaning, disinfection and overnight storage of contact lenses
  Other Names: CLEAR CARE® PLUS
Device: Habitual Multi-Purpose Contact Lens Solution
Device: Habitual Contact Lenses — Participant's habitual contact lens brand worn in a daily wear modality for 30 days.

SUMMARY:
The purpose of this study is to evaluate CLEAR CARE® PLUS (CCP) compared to non-HYDRAGLYDE® multi-purpose contact lens solutions in presbyopes currently wearing soft contact lenses and experiencing symptoms of dryness.

ELIGIBILITY:
Inclusion Criteria:

* Must sign an informed consent document;
* Current adapted two-week/monthly replacement soft contact lens wearers (at least 2 months) with symptoms of contact lens induced dryness;
* Near spectacle add of +0.50 or greater;
* Best corrected visual acuity (BCVA) to 20/30 or better in each eye at distance;
* Willing to wear lenses for a minimum of 5 days per week, 6 hours per day, and attend all study visits;
* Currently (at least 2 months) using a non-HYDRAGLYDE® containing multi-purpose solution (OPTI-FREE® PureMoist® is excluded) to care for lenses;
* Use of digital devices (eg, smart phone, tablet, laptop computer, or desktop computer) for 20 consecutive minutes at least twice a week and willing to continue the same pattern for the duration of the study;
* Other protocol-specific inclusion criteria may apply.

Exclusion Criteria:

* Extended wear contact lens wearer (sleeps in lenses 1 or more nights per week);
* Any anterior segment infection, inflammation, disease, or abnormality that contraindicates contact lens wear as determined by the investigator;
* Any use of systemic or ocular medications for which contact lens wear could be contraindicated, as determined by the investigator, including use of any topical ocular medications that would require instillation during contact lens wear;
* Monocular (only 1 eye with functional vision) or fit with only 1 lens;
* Known sensitivity to any ingredients in CLEAR CARE® PLUS (CCP);
* Prior refractive surgery;
* History of herpetic keratitis, ocular surgery, or irregular cornea;
* Pathological dry eye that precludes contact lens wear;
* Use of mechanical eyelid therapy or eyelid scrubs within 14 days before Visit 1 and not willing to discontinue during the study;
* Participation in any clinical study within 30 days of Visit 1;
* Currently using or have not discontinued Restasis®, Xiidra® or a topical steroid within the past 7 days;
* Other protocol-specific exclusion criteria may apply.

Ages: 45 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 126 (Actual)
Dates: Start 2016-12-13 (Actual); Primary Completion 2017-03-24 (Actual); Study Completion 2017-03-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Project Manager, CPM, Study Director — Alcon, A Novartis Division

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from 9 study centers located in the United States.
Pre-assignment Details: Of the 126 enrolled, 5 subjects were exited as screen failures prior to randomization. This reporting group includes all randomized subjects (121).
Groups:
- CCP/HMPS: 3% hydrogen peroxide solution with HydraGlyde® Moisture Matrix contact lens solution (CCP) in Period 1, followed by subject's habitual multi-purpose contact lens solution (HMPS) in Period 2. Each product used daily per packaging instructions with subject's habitual contact lenses for approximately 30 cleaning and disinfection cycles.
- HMPS/CCP: Subject's habitual multi-purpose contact lens solution in Period 1, followed by 3% hydrogen peroxide solution with HydraGlyde® Moisture Matrix contact lens solution in Period 2. Each product used daily per packaging instructions with subject's habitual contact lenses for approximately 30 cleaning and disinfection cycles.
Period: Period 1, First 30 Days of Wear
Arm/Group | CCP/HMPS | HMPS/CCP
Started | 67 | 54
Completed | 64 | 52
Not Completed | 3 | 2
Not completed — Adverse Event | 0 | 1
Not completed — Lost to Follow-up | 1 | 1
Not completed — Protocol Violation | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0
Period: Period 2, Second 30 Days of Wear
Arm/Group | CCP/HMPS | HMPS/CCP
Started | 64 | 52
Completed | 62 | 52
Not Completed | 2 | 0
Not completed — Protocol Violation | 2 | 0

BASELINE CHARACTERISTICS:
Population: This analysis set includes all randomized subjects who were exposed to at least one of the study lens care products evaluated in this study (Full Analysis Set).
Groups:
- Overall: 3% hydrogen peroxide solution with HydraGlyde® Moisture Matrix and subject's HMPS used during Period 1 and Period 2 in a crossover assignment.
Arm/Group | Overall
Number analyzed (Participants) | 121
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.5 (5.54)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 104
  Male | 17
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 119
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 16
  White | 103
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Contact Lens Dry Eye Questionnaire-8 (CLDEQ-8) Score at Day 30
Description: CLDEQ-8 score (assessment of contact lens discomfort) was obtained by adding the numerical responses to each of 8 items. Individual scales ranged from 0-4, 0-5, and 1-6, with a resultant overall score from 1 minimum to 37 maximum. A lower CLDEQ-8 score indicates less frequent or less intense symptoms.
Time Frame: Day 30, each product
Population: Full Analysis Set with non-missing responses
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- CLEAR CARE PLUS: 3% hydrogen peroxide solution with HydraGlyde® Moisture Matrix contact lens solution used daily with subject's habitual contact lenses for approximately 30 cleaning and disinfection cycles.
- HMPS: Subject's habitual multi-purpose contact lens solution used daily with subject's habitual contact lenses for approximately 30 cleaning and disinfection cycles.
Arm/Group | CLEAR CARE PLUS | HMPS
Number analyzed (Participants) | 114 | 117
units on a scale | 12.6 (7.19) | 14.8 (7.99)
Statistical Analysis 1: Comparison: CLEAR CARE PLUS vs HMPS; Test type: Superiority; p = 0.0073, Mixed Models Analysis

ADVERSE EVENTS:
Time Frame: Day 1 through study completion, an average of 60 days
Description: An AE was defined as any untoward medical occurrence, unintended disease or injury, or untoward clinical signs in subjects, users, or other persons, whether or not related to the investigational medical device. AEs were obtained through solicited and spontaneous comments from subjects and through observations by the Investigator.
Groups:
- CLEAR CARE PLUS: All subjects exposed to CCP contact lens solution
- HMPS: All subjects exposed to habitual multi-purpose contact lens solution
Arm/Group | CLEAR CARE PLUS | HMPS
All-Cause Mortality (participants affected / at risk) | 0/121 | 0/121
Serious Adverse Events (participants affected / at risk) | 0/121 | 1/121
Other Adverse Events (participants affected / at risk) | 0/121 | 0/121
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | CLEAR CARE PLUS (N=121) | HMPS (N=121)
Colorectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor reserves the right of prior review of any publication or presentation of information related to the study.

DOCUMENTS (2):
  • Study Protocol (2016-12-20): https://cdn.clinicaltrials.gov/large-docs/33/NCT02965833/Prot_000.pdf
  • Statistical Analysis Plan (2015-03-16): https://cdn.clinicaltrials.gov/large-docs/33/NCT02965833/SAP_001.pdf